CLINICAL TRIAL: NCT02521896
Title: Vado™ Steerable Sheath System; A Safety and Performance Study to Evaluate Access to the Pulmonary Veins in the Treatment of Paroxysmal and Persistent Atrial Fibrillation
Brief Title: Safety and Performance Study to Evaluate Access to Pulmonary Veins for Treatment of Paroxysmal AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kalila Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP1-001
Record Dates: First submitted 2015-08-06; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Steerable sheath for intracardiac access (Experimental): Vado Steerable sheath system consisting of a dilator and steerable sheath for left atrial access, positioning of ablation catheters and placement of mapping and ablation catheters for circumferential ablation
  Interventions: Device: Steerable Sheath System

INTERVENTIONS:
Device: Steerable Sheath System — The Vado™ Steerable Sheath consists of a dilator and steerable sheath which are designed to provide intracardiac access and flexible catheter positioning in the cardiac anatomy.
  Other Names: Vado Steerable Sheath

SUMMARY:
The study is intended to assess the safety and performance of the Vado™ Steerable Sheath in facilitating ease of access to the pulmonary veins (PV) for the treatment of paroxysmal atrial fibrillation and persistent atrial fibrillation (AF). The study will be a prospective, single-center, non-randomized investigation.

DETAILED DESCRIPTION:
The design for this study involves the sequential enrollment of patients with documented paroxysmal atrial fibrillation who have had two (2) or more AF episodes for at least 30 seconds in length within six (6) months prior to enrollment. Target population shall be selected from the treatable AF population that meets both inclusion/exclusion criteria.It is intended that the Vado Steerable Sheath will be used as part of standard clinical workflow procedures, with no procedural deviations relative to other procedures requiring steerable sheaths. Individual subjects will be studied during mapping and ablation procedures and followed until release from hospital post procedure per institutional standard of care.

ELIGIBILITY:
Inclusion Criteria:

* suitable candidate for intra-cardiac mapping for arrhythmias with documented PAF defined by HRS Criteria.
* Eighteen to Eighty years of age
* Signed informed consent

Exclusion Criteria:

* Intracardiac thrombus, tumor or other abnormality that precludes catheter introduction and placement
* Severe cerebrovascular disease or history of cerebrovascular event within one (1) month
* Patients with severely impaired kidney function as measured by a Cockcroft-Gault Glomerular Filtration Rate (GFR) 3 with a GFR < 29.
* Active gastrointestinal bleeding, infection or fever (> 100.5/38C)
* Severe co morbidity or Short life expectancy (<1 year) due to other illnesses such as cancer, pulmonary, hepatic or renal disease
* Structural heart disease of clinical significance including

  * Symptoms of congestive heart failure including, but not limited to, NYHA Class III or IV CHF and/or documented ejection fraction < 40% measured by acceptable cardiac testing
  * Stable/unstable angina or ongoing myocardial ischemia
  * Myocardial infarction (MI) within three months of enrollment
  * Aortic or mitral valve disease > Grade II
  * Congenital heart disease (not including ASD or PFO without a right to left shunt) where the underlying abnormality increases the risk of an ablative procedure
* Enrollment in any other ongoing arrhythmia study protocol
* Any ventricular tachyarrhythmia currently being treated where the arrhythmia or the management may interfere with this study
* Active infection or sepsis
* Female patient is pregnant or lactating
* Untreatable allergy to contrast media
* Any diagnosis of atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or any other reversible or non-cardiovascular causes
* History of blood clotting (bleeding or thrombotic) abnormalities
* Known sensitivities to heparin or warfarin
* Severe COPD (identified by an FEV1 <1)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Absence of adverse device related events at release from hospital post procedure per institutional standard of care | Procedure through 7 day clinical follow up
  Steerability and positioning to facilitate catheter placement

SECONDARY OUTCOMES:
Hemostasis and Visibility of the steerable sheath | Procedure through 7 day clinical follow up
  Safe event free insertion of the steerable sheath system in the femoral vein

CONTACTS AND LOCATIONS:
Overall Officials: Ian Crozier, MD, Principal Investigator — Christchurch Hospital; Matthew Daly, MD, Principal Investigator — Christchurch Hospital

REFERENCES:
- [Background] Piorkowski C, Eitel C, Rolf S, Bode K, Sommer P, Gaspar T, Kircher S, Wetzel U, Parwani AS, Boldt LH, Mende M, Bollmann A, Husser D, Dagres N, Esato M, Arya A, Haverkamp W, Hindricks G. Steerable versus nonsteerable sheath technology in atrial fibrillation ablation: a prospective, randomized study. Circ Arrhythm Electrophysiol. 2011 Apr;4(2):157-65. doi: 10.1161/CIRCEP.110.957761. Epub 2011 Jan 19. PMID 21248246